CLINICAL TRIAL: NCT04227938
Title: An Open-label Study of ALPN-101 in Steroid-resistant or Steroid-refractory Acute Graft Versus Host Disease (aGVHD)
Brief Title: ALPN-101 in Steroid-resistant or Steroid-refractory Acute GVHD
Acronym: Balance
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Change in sponsor strategy
Sponsor: Alpine Immune Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AIS-A02
Record Dates: First submitted 2020-01-06; First posted 2020-01-14 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2020-08

CONDITIONS: Graft Vs Host Disease
Keywords: steroid-resistant acute graft versus host disease; steroid-refractory acute graft versus host disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — ALPN-101

STUDY DESIGN:
Intervention Model Description: A single dose of ALPN-101 will be administered via intravenous (IV) infusion. Multiple, ascending dose levels will be evaluated in cohorts of 3-6 subjects in Part A. In Part B, a single dose level-as identified in Part A-is planned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ALPN-101 (Experimental): All subjects will receive a single dose of ALPN-101. In Part A, ascending dose levels of ALPN-101 will be evaluated. In Part B, a single dose level of ALPN-101-as identified in Part A-will be evaluated.
  Interventions: Drug: ALPN-101

INTERVENTIONS:
Drug: ALPN-101 — A single dose of ALPN-101 will be administered via intravenous infusion.

SUMMARY:
The Balance study will assess the safety, tolerability, and efficacy of an investigational drug called ALPN-101 in adults with steroid-resistant or steroid-refractory acute graft versus host disease (aGVHD).

DETAILED DESCRIPTION:
AIS-A02 is a Phase 1b open-label study of ALPN-101 administered to adult subjects with steroid-resistant or steroid-refractory acute graft versus host disease (aGVHD).

It will be conducted at approximately 10 US sites. Up to 72 subjects will be enrolled in Part A (dose escalation) and up to 25 subjects will be enrolled in Part B (dose expansion).

In each Part, safety and efficacy assessments will be performed throughout the dosing and follow-up periods, and multiple PK and PD samples will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Status post first allogeneic stem cell transplantation (allo-SCT) from any donor source using any conditioning regimen.
3. Grade Ⅱ-Ⅳ acute GVHD per Mount Sinai Acute GVHD international Consortium (MAGIC) criteria.
4. Corticosteroid resistant or refractory as defined as any of the following:

   1. Progression of aGVHD within 5 days following initiation of treatment with ≥ 2 mg/kg/day of prednisone or equivalent;
   2. Failure to improve within 7 days following initiation of treatment with ≥ 2 mg/kg/day of prednisone or equivalent; or
   3. Incomplete response (failure to achieve Complete Response) after 28 days of immunosuppressive treatment including steroids (treatment with ≥ 2 mg/kg/day of prednisone or equivalent).
5. Must agree to use appropriate contraception.
6. Female subjects must not be pregnant or breastfeeding.

   In addition, the following criteria must be met prior to dosing with ALPN-101 on Day 1:
7. Karnofsky performance score ≥ 40.
8. No evidence of an active, uncontrolled bacterial, viral, or fungal infection.

Exclusion Criteria:

1. Current veno-occlusive disease, or current treatment with dialysis or mechanical ventilation associated with GVHD.
2. Prior donor lymphocyte infusion (DLI).
3. Receipt of any live vaccine within 4 weeks of ALPN-101 dosing.
4. Presence of any active malignant disease.
5. Corticosteroid therapy at doses > 1 mg/kg/day prednisone or equivalent for indications other than GVHD ≤ 7 days p ALPN-101 dosing.
6. Treatment with any of the following ≤ 2 weeks prior to ALPN-101 dosing: targeted inhibitors of the CD28/CD80/86 pathway (e.g. abatacept, belatacept), targeted inhibitors of the ICOS/ICOSL pathway
7. Initiation of treatment with salvage therapy < 2 days prior to ALPN-101 dosing. Concurrent salvage therapy that is intended to be continued must be at a stable dose for ≥ 2 days prior to ALPN-101 dosing.
8. Treatment for aGVHD with adoptive cell therapy, investigational agents, devices, or procedures ≤ 2 weeks or 5 half-lives-whichever is greater-prior to ALPN-101 dosing, unless approved by the medical monitor and sponsor; prior treatment with mesenchymal stem cells is permitted.
9. Known allergies, hypersensitivity, or intolerance to study drug, excipients, or similar compounds.
10. Any medical complications or conditions that would, in the investigator's judgment, interfere with full participation in the study, including administration of study drug and attending required study visits; pose a significant risk to the participant; or interfere with interpretation of study data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2020-05-21 (Actual); Study Completion 2020-05-21 (Actual)

PRIMARY OUTCOMES:
Adverse events | From study Day 1 (dosing of ALPN-101) until Day 29
  The incidence, severity, and seriousness of AEs, including dose-limiting toxicities, assessed by CTCAE

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | From study Day 1 (dosing of ALPN-101) until the date of best response, assessed up to 36 months
  Assessed by MAGIC criteria
Duration of Response (DOR) | From the date of best response until disease progression, assessed up to 36 months
Failure-free survival (FFS) | From study Day 1 (dosing of ALPN-101) until relapse, initiation of new systemic therapy, or non-relapse mortality; assessed up to 36 months
Event-free survival (EFS) | From study Day 1 (dosing of ALPN-101) until disease (aGVHD)-related event or death due to any cause, assessed up to 36 months
Non-relapse mortality (NRM) | From study Day 1 (dosing of ALPN-101) until progression or death due to any cause without prior progression, assessed up to 36 months
Malignancy relapse/progression (MR) | From study Day 1 (dosing of ALPN-101) until the date of relapse/progression of the primary malignancy, assessed up to 36 months
Overall survival (OS) | From study Day 1 (dosing of ALPN-101) until death due to any cause, assessed up to 36 months
Time to maximum observed concentration (tmax) of ALPN-101 | From study Day 1 (dosing of ALPN-101) until Day 29
Maximum observed concentration (Cmax) of ALPN-101 | From study Day 1 (dosing of ALPN-101) until Day 29
Area under the concentration-time curve (AUC) of ALPN-101 | From study Day 1 (dosing of ALPN-101) until Day 29

CONTACTS AND LOCATIONS:
Overall Officials: Jan Hillson, MD, Study Director — Alpine Immune Sciences, Inc.
Locations (4):
- United States (4):
  - University of Miami, Miami, Florida
  - University of Kansas Hospital, Kansas City, Kansas
  - Sarah Cannon Center for Blood Cancer, Nashville, Tennessee
  - St. David's South Austin medical Center, Austin, Texas

IPD SHARING:
Plan to Share IPD: No